CLINICAL TRIAL: NCT01126658
Title: Evaluation of the Intracranial Volume Pressure Relationship in Increased Intracranial Pressure Patients by a Mathematic Manner
Brief Title: Evaluation the Intracranial Volume Pressure Response in Increased Intracranial Pressure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Chang Gung Memorial Hospital, Chang Gung Medical Research Council
Other Study IDs: CMRPG 371581
Record Dates: First submitted 2010-05-18; First posted 2010-05-20 (Estimated); Last update posted 2010-05-24 (Estimated); Status verified 2010-05

CONDITIONS: Brain Injury; Intracranial Hypertension
Keywords: pressure-volume curve; intracranial pressure; volume pressure response; pressure-volume relationship; mathematical model
MeSH Terms: conditions — Brain Injuries; Intracranial Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- All subjects act as their own contral
  Interventions: Other: drainage of cerebrospinal fluid (CSF)

INTERVENTIONS:
Other: drainage of cerebrospinal fluid (CSF) — Once the ICP exceed 20-25 mmHg, 1 ml of CSF was withdrawn from EVD and the corresponding change of ICP value was recorded. The withdrawn drainage of CSF continued until the final ICP value declined to 10 mmHg.

SUMMARY:
The purpose of this study is to discover a mathematic equation to express the intracranial pressure-volume (P-V) curve and a single indicator to reflect the status of the curve.

DETAILED DESCRIPTION:
Monitoring of intracranial pressure (ICP) has been used in the management of patients with increased ICP, or in whom increased ICP was suspected. ICP depends on the relative constancy of total volume inside the skull, comprising cerebrospinal fluid (CSF), blood, and brain tissue. The changes of CSF volume affect the ventricular fluid pressure and defined it as volume pressure response (VPR). The shape or curve of the intracranial volume-pressure (V-P) relationship is well known in daily neurosurgical practice. If the P-V curve can be expressed by mathematic manner, then there should be an indicator to reflect the status of the curve. This study is conducted in order to understand the difference of each P-V curve in patients with increased intracranial pressure. The individual VPR values have been tested with three mathematical models (linear, parabolic and exponential regression equation).

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe brain damage
* Underwent bilateral external ventricular drainage (EVD)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: over 30 patients with severe brain injury and underwent bilateral external ventricular drainage in situ.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-02 (Actual); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
intracranial pressure | one minute.
  The ICP values were obtained from the bedside ICU monitor. Once the ICP values exceed 20-25 mmHg, 1 ml of CSF was withdrawn from EVD and the corresponding change of ICP value was recorded. The withdrawn drainage of CSF continued until the final ICP value declined to 10 mmHg and the whole drainage procedure was completed within one minute.

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Tseng Lee, MD, Study Chair — Department of Neurosurgery,Chang Gung Memorial Hospital; Hung-Yi Lai, MD, Principal Investigator — Department of Neurosurgery,Chang Gung Memorial Hospital
Locations (1):
- Department of Neurosurgery,Chang Gung Memorial Hospital, Taoyuan District, Taiwan

REFERENCES:
- [Derived] Lai HY, Lee CY, Hsu HH, Lee ST. The intracranial volume pressure response in increased intracranial pressure patients: Part 1. Calculation of the volume pressure indicator. Acta Neurochir (Wien). 2012 Dec;154(12):2271-5; discussion 2275. doi: 10.1007/s00701-010-0765-8. Epub 2010 Aug 18. PMID 20714759